CLINICAL TRIAL: NCT05093348
Title: Pseudonymised Single Site Investigation Into Unique Patient Data Acquisition Using Anterior Segment Optical Coherence Tomography for the Digital Design and Manufacture of Ocular Prosthesis and Randomised Crossover Trial of Analogue Versus Digital Ocular Prosthesis
Brief Title: Click2Print Artificial Eyes
Acronym: Click2Print
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SAGM1006
Record Dates: First submitted 2021-08-11; First posted 2021-10-26 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Enucleated; Eye; Evisceration; Traumatic, Eye
Keywords: Enucleated; Artificial eye; Prosthesis; Eviscerated

STUDY DESIGN:
Intervention Model Description: Pseudonymised single site investigation randomised crossover trial
Who Masked: Participant, Investigator
Masking Description: Demographics will be such that the data subject cannot be identified. It will not be possible to mask the ocularist, data manager or the trial manager. Every effort will be made to mask the patient and investigators from knowing which type of prosthesis is being worn during the trial. However, due to the differing methods of manufacture of a digital artificial eye compared to the traditional artificial eye, upon close inspection, it may be possible to denote differences in the cosmetic appearance. Should the participant ask or comment on which type of artificial eye they are wearing to the ocularist or research member then a scripted response will be provided.
  The trial statistician who is analysing trial data will be masked until primary analysis is completed. Un-masking of the ocular prosthesis will occur after confirmation of primary analysis has been performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Click2Print digital Artificial Eye (Active Comparator): Supply and fit a digitally designed and manufactured ocular prosthesis for four months in comparison to the current hand-made ocular prosthesis in a cross over trial
  Interventions: Device: Click2Print artificial eye
- Current hand made artificial eye (Active Comparator): Wear the hand-made artificial eye for four months and compare to the digitally design ed and manufactured artificial eye
  Interventions: Device: Hand-made artificial eye

INTERVENTIONS:
Device: Click2Print artificial eye — Digitally designed and manufactured ocular prosthesis
  Arms: Click2Print digital Artificial Eye
Device: Hand-made artificial eye — Hand-made artificial eye
  Arms: Current hand made artificial eye

SUMMARY:
To undertake a randomised crossover trial in human subjects the Click2Print ocular prosthesis versus an analogue ocular prosthesis demonstrating non-inferiority in the assessment of ocular prosthesis motility, cosmesis, fit and function, comfort, mucous discharge and benefits of use in daily life in 40 data subjects (Crossover Trial).

DETAILED DESCRIPTION:
For this project, the investigators will conduct a randomised controlled crossover trial comparing the efficacy, safety and performance of the Click2Print ocular prosthesis versus the handmade analogue ocular prosthesis.

A non-invasive image is taken on an anterior segment optical coherence tomography device (AS-OCT), which captures data subject data of the anophthalmic socket so that the anatomy of the anterior orbit can be outlined. At the same sitting the data of the fellow eye is captured by taking an AS-OCT of the volume of the cornea and iris.

Simultaneously a colour calibrated image of the fellow eye is captured. This unique data will serve as a template for the design of the bespoke Click2Print ocular prosthesis. The investigators anticipate that the Click2Print ocular prosthesis will not be inferior in fit and function to the handmade analogue ocular prosthesis. The Click2Print ocular prosthesis is also expected to match the analogue ocular prosthesis in the objective measures of prosthesis motility and cosmesis and that there will be no adverse events in terms of the socket and general health.

Statistical methodology and analysis:

The study design is a randomised, crossover trial of Click2Print ocular prosthesis versus analogue ocular prosthesis. The methods will include a non-inferiority comparison of ocular motility between the two prosthesis types, and a standard comparison of subjective outcomes including: cosmesis, comfort, and durability of colour and structure. The analysis will include the development of a non-inferiority margin for the comparison of motility, non-parametric significance tests for questionnaire data, and parametric significance tests for volume data. The alpha level is 0.05 and superiority significance tests will be two-tailed.

Evaluation of clinical data that are relevant to the proposed clinical investigation.

The data will be statistically analysed to determine if a Click2Print ocular prosthesis is non inferior in motility and in comparison, to an analogue ocular prosthesis. Cosmesis will be assessed by standard comparison of subjective outcomes.

Data subjects will be requested to complete a general ocular prosthesis questionnaire. The questionnaire will help to evaluate how a Click2Print ocular prosthesis compares to the current analogue ocular prosthesis. Topics covered in the questionnaire will be:

* Cosmesis
* Fit and function
* Comfort
* Motility
* Mucoid discharge
* Benefits

Risk to benefit rationale.

The result of the risk management process is that the residual risks, as identified in the risk analysis, as well as risk(s) to the subject associated with the clinical procedure are outweighed by the anticipated benefits to the subjects.

Procedures to be taken in case of adverse events:

All adverse events and serious adverse events will be recorded in the medical records and case report form. All serious adverse events will be reported to the sponsor.

Description of the measures taken to minimize or avoid bias, including randomization and blinding/masking.

Data subjects enrolled in the clinical investigation will be allocated a study number. Randomisation allocation of first ocular prosthesis wear by patient will be assigned, using allocation concealment, against consecutive Study IDs. After 4 months, patient will crossover to receive the alternative prosthesis. The randomisation list will be generated centrally using random permutated blocks of varying sizes in STATA statistical software. Seed number will be recorded for future reference in the original randomisation list.

Demographics will be such that the data subject cannot be identified. Every effort will be made to mask the patient and investigators from knowing which type of prosthesis is being worn during the trial.

The trial statistician who is analysing trial data will be masked until primary analysis is completed.

Methods and timing for assessing, recording, and analysing variables.

* General Ocular Prosthesis Questionnaire visits 3,4,5 and 6
* Cosmesis assessment visit 2 and visit 4
* Motility assessments visits 2, 3, 4 and 5

Monitoring plan

Case Report Forms will be completed by the investigator and/or delegates within 2 working days of the study visit. All data from the examinations and investigations will be transferred to media provided by the sponsor and collected at the time of collection.

Moorfields Eye Hospital NHS Foundation Trust, the sponsor, will perform interim monitoring visits. These will be undertaken by an independent monitor contracted with Moorfields.

Trial Management Group(TMG)

The TMG will monitor all aspects of the conduct and progress of the trial, ensure that protocol is adhered to and take appropriate action to safeguard participants and the quality of the trial itself. The group will meet to discuss any issues with data quality and any concerns will be discussed at the trial steering committee

Independent Data Monitoring Committee (IDMC)

An IDMC will monitor the trial progress and patient safety data, at intervals, while the clinical trial is ongoing. The IDMC will make recommendations to the TSC regarding continuation, stopping or any modification to the trial.

Trial Steering Committee (TSC)

A TSC will be set up to provide the overall supervision of the trial and ensure that it is being conducted in accordance with the principles of good clinical practice and the relevant regulations. The TSC will have an independent chair and include members (including one lay member) who are independent of the investigators, their employing organisations, funders and sponsors. The TSC will agree the trial protocol and any protocol amendments, monitor trial progress, monitor trial conduct and advise on scientific credibility. The TSC will consider and act, as appropriate, upon the recommendations of the IDMC or equivalent and ultimately carries the responsibility for deciding whether a trial needs to be stopped on grounds of safety or efficacy.

Confidentiality All data will be handled in accordance with the General Data Protection Regulation (GDPR) and United Kingdom Data Protection Act 2018. The case report forms will not bear the subject's name or other personal identifiable data. The trial identification number will be used for identification. Subjects will be assigned a trial identification number by the study site sequentially starting with {01} upon enrolment into the study. The study site will maintain a master Subject Identification Log.

Record keeping and archiving Archiving will be authorised by the Sponsor following submission of the end of study report. Chief Investigators are responsible for the secure archiving of essential trial documents as per trust policy. All essential documents will be archived in line with the sponsor archiving procedure after completion of trial. Destruction of essential documents will require authorisation from the Sponsor.

Statistical Analysis Plan:

The statistical analysis will be completed by Dr. Andrew W. Stacey. The analysis will be completed using the R Statistical Environment software. The following analyses will be completed:

* Demographic data will be listed as descriptive data only, there is no concern for difference between groups in this cross-over design, and therefore no comparison between groups is necessary.
* Design: The comparison of ocular prosthesis motility is designed as a non-inferiority study. Therefore, the null hypothesis is taken to be that the new Click2Print ocular prosthesis is inferior to the standard analogue prosthesis. If the null hypothesis is rejected, the trial demonstrates non-inferiority of the Click2Print ocular prosthesis device (Device 1) compared to the analogue ocular prosthesis.
* Ocular Motility: Ocular motility measurements will be calculated in four directions of gaze in each eye (upgaze, downgaze, adduction and abduction). For each direction of excursion, a ratio will be calculated as follows: excursion of the analogue ocular prosthesis divided by excursion of the Click2Print ocular prosthesis. When the ratio equal "1", the two measurements are equal. A number greater than 1 indicates better excursion in the analogue ocular prosthesis. A number less than 1 indicates better excursion in the Click2Print ocular prosthesis. A 95% confidence interval will be calculated around this ratio using data from all subjects in the trial. The confidence interval will be compared to the non-inferiority margin.
* Non-inferiority margin for excursion: There is little published research or a priori data for comparison of different ocular prosthesis options. Pilot data from this study demonstrated mean excursions of the analogue implant to be: adduction: 1.6mm, abduction: 1.5mm, upgaze: 4.0mm, downgaze: 2.1mm. It was determined that a difference of greater than 25% motility would be necessary to see a clinically appreciable decrease between the Click2Print ocular prosthesis and the analogue ocular prosthesis. The non-inferiority margin for excursion was set at 25% of the excursion of the analogue implant. If the upper limit of the 95% confidence interval of the ratio of excursions is less than 1.25, the null hypothesis will be rejected and the Click2Print ocular prosthesis prothesis will be demonstrated to be non-inferior.
* A Total Motility Score (TMS)will be calculated by adding all four directions of gaze together. This will be compared in similar fashion with a 95% confidence interval as described above and with a similar non-inferiority margin.
* Cosmesis Assessment: Data from the cosmesis assessment represent ordinal data. Due to the subjective nature of these data, the results will be analysed with standard statistical tests of superiority. These data will be analysed using non-parametric tests, specifically Mann-Whitney. Data subject subjective responses will be compared between groups.
* Each ocular prosthesis will undergo volumetric analysis as described previously. The volume will be calculated for the analogue ocular prosthesis and the Click2Print ocular prosthesis at the beginning and end of the trial period. The before and after volume data will be compared to determine if any change in volume occurred while the device was being worn by the data subject. These continuous data will be compared with Student T-tests.
* Each ocular prosthesis will undergo a colorimetric analysis after the trial period. A photograph will be taken, as previously described, at the beginning and end of each trial period. The "before" and "after" photos will be graded by two separate, independent graders. The graders will be asked to compare the colour of the "before" photo to the colour of the "after" photo. The graders will be given two options for each data subject and each ocular prosthesis type: "equal" or "not equal". Interrater reliability will be calculated to verify reliability. The rate of "equal" and "not equal" results for both prostheses will be compared using Fisher-exact tests.
* General Ocular Prosthesis Questionnaire: This is a 5-point Likert-type scale. The analysis will be similar to the cosmesis assessment with direct comparison of groups using non-parametric statistical tests (Mann-Whitney).
* Data subject Diary: Data from the data subject diary will be qualitative, these data will be analysed only with prose and descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and over
* Adults with surgery to remove one eye with at least 1-year follow-up
* Able to give consent and understand the study
* Able to cooperate by following instructions

Exclusion Criteria:

* - Adults with surgery to remove one eye with less than 1-year follow-up.
* Concurrent socket pathology (Socket infection or exposure).
* Giant papillary conjunctivitis.
* Presence of ocular motility disorders on either side of the face, muscle restrictive disorders, previous trauma, idiopathic orbital inflammatory disease and neurological disorders (cranial neuropathies, multiple sclerosis).
* Data subjects unable to understand the study and unable to give informed consent.
* Data subjects considered vulnerable.
* Ongoing participation in another clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2023-07-16 (Actual); Study Completion 2023-07-16 (Actual)

PRIMARY OUTCOMES:
Comparison of prosthesis motility utilising an excursion assessment to prove non-inferiority of the digital ocular prosthesis | 8 months
  Each subject will use two different ocular prostheses for an extended period of time and the motility of each will be compared. Each ocular prosthesis will be worn for 4 months. Motility will be assessed at the beginning and after 3 month period of wear for each prosthesis. Motility will be measured by assessing the ocular prosthesis excursion in four angles of gaze. The distance from straight ahead gaze compared to left, right, up and down gaze will be measured in millimetres and recorded on the case report form. These measurements will then be used to compute a total motility score. The data subject will cross-over to wearing the comparator type prosthesis and the motility assessment will be repeated at the beginning and after three month period. The total motility scores of type 1 and type 2 prostheses will then be compared to determine if the digital ocular prosthesis motility is non-inferior to the gold-standard handmade prosthesis.

CONTACTS AND LOCATIONS:
Overall Officials: Mandeep Sagoo, Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust
Locations (1):
- Moorfields Eye Hospital NHS Foundation Trust, 162 City Road, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All participant data will remain within the sponsor organisation